CLINICAL TRIAL: NCT03002623
Title: A Phase II Trial of CUDC-907 in Patients With Metastatic and Locally Advanced Thyroid Cancer
Brief Title: CUDC-907 Treatment in People With Metastatic and Locally Advanced Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed because investigator left the National Institutes of Health.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170029; 17-C-0029
Record Dates: First submitted 2016-12-22; First posted 2016-12-26 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Thyroid Neoplasms; Poorly Differentiated and Undifferentiated Thyroid Cancer; Differentiated Thyroid Cancer
Keywords: Dual Inhibitor of HDAC and P13K Signaling; HDAC2; EGFR/RAS/RAF/MEK/ERK Signaling Pathway Inhibition
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Carcinoma, Anaplastic | interventions — CUDC-907

STUDY DESIGN:
Intervention Model Description: This is a single group assignment. All patients regardless of subtype of thyroid cancer received one single treatment and follow up plan with option to continue the treatment when scan was negative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): CUDC-907 for thyroid cancer
  Interventions: Drug: CUDC-907

INTERVENTIONS:
Drug: CUDC-907 — 60 mg (2 capsules of 30 mg capsules) will be given orally once a day 5 days on and 2 days off.

SUMMARY:
Background:

The thyroid is a gland at the base of the throat. Thyroid cancer is a disease that people get when abnormal cells begin to grow in this gland. Researchers believe a new drug called CUDC-907 may be able to help people with thyroid cancer that has spread or has gotten worse.

Objective:

To see if CUDC-907 will shrink tumors in people with advanced thyroid cancer.

Eligibility:

People at least 18 years old who have been diagnosed with locally advanced and metastatic thyroid cancer.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Electrocardiogram (ECG) heart test.

Review of their symptoms and how they perform normal activities

A scan will be performed. Some will have a computed tomographic scan (CT) that takes pictures of the body using a small amount of radiation. Some will have magnetic resonance imaging (MRI) that uses a magnetic field to take pictures.

Bone scan (some participants)

Fludeoxyglucose (FDG) positron emission tomography (PET) scan to produce a tumor image.

A sample of their tumor from a previous surgery. They may have a biopsy of their tumor if a tumor sample is not available from a previous surgery.

Participants will be given CUDC-907 in tablet form. They will take it by mouth once a day for 5 days, then take 2 days off, each week.

While taking the study drug, participants will have study visits that repeat the screening tests.

After they stop treatment, participants will have 3 follow-up visits over a year. They will repeat some tests. Then participants will be contacted by phone or e-mail every 6 months....

DETAILED DESCRIPTION:
Background:

* There are no standard or effective systemic therapies for metastatic or locally advanced poorly differentiated and undifferentiated thyroid cancer.
* Poorly differentiated and undifferentiated thyroid cancer are aggressive, with high mortality.
* CUDC-907 is a first-in-class dual inhibitor of histone deacetylase (HDAC) and PI3K signaling.
* Approximately 80% of poorly differentiated and undifferentiated thyroid cancers have driver mutations in the PI3K/AKT pathway or activation of the pathway.
* HDAC2 is upregulated in poorly differentiated and undifferentiated thyroid cancer, and aggressive variants of differentiated thyroid cancer, and CUDC-907 treatment reduces HDAC2 levels in thyroid cancer cells.
* CUDC-907 inhibits thyroid cancer cell growth, invasion and migration in vitro.
* In addition to inhibiting the PI3K/AKT signaling pathway, CUDC-907 inhibits the EGFR/RAS/RAF/MEK/ERK signaling pathway, which is also activated in poorly differentiated and undifferentiated thyroid cancer.
* CUDC-907 inhibits growth and metastases in a mouse model of metastatic thyroid cancer.
* We hypothesize that CUDC-907 will cause cancer regression in patients with metastatic and locally advanced poorly differentiated and undifferentiated thyroid cancer, and aggressive variants of differentiated thyroid cancer.

Objective:

-To determine response to CUDC-907 treatment by Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with locally advanced and metastatic poorly differentiated and undifferentiated thyroid cancer, and aggressive variants of differentiated thyroid cancer.

Eligibility:

* Age greater than or equal to 18 years
* Thyroid cancer that is refractory to or relapsed after standard treatment.
* Aggressive thyroid cancer confirmed on histology or cytologic analysis.
* Measurable disease.
* Last dose of chemotherapy or last radiotherapy treatment more than 4 weeks prior to starting treatment with this protocol, except for subjects with anaplastic/undifferentiated thyroid cancer who may enroll immediately after discontinuation of previous therapy.

Design:

* Open label, phase II trial to determine response to CUDC-907 treatment.
* Patients will be given 60 mg of CUDC-907 orally for 5 consecutive days followed by 2 days off (5/2 schedule).
* One cycle is 21 days. Patients may continue on treatment if there is no disease progression.
* Initial anatomic and functional imaging will be performed at enrollment and after 2 cycles of treatment. Thereafter, anatomic imaging will be performed every two cycles of treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects greater than or equal to 18 years of age.
* Thyroid cancer histology or cytology that is aggressive (anaplastic/undifferentiated thyroid cancer, poorly differentiated thyroid cancer, Hurthle cell carcinoma, tall-cell variant of papillary thyroid cancer, sclerosing variant of papillary thyroid cancer).
* Measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Absolute neutrophil count greater than or equal to 1,000/microL
* Platelets greater than or equal to 75,000/microL
* Creatinine less than or equal to 1.5 times upper limit of normal (ULN) or creatinine clearance > 60ml for patients with creatinine levels 1.5 times above institutional ULN (calculated based on age, weight and sex
* Total bilirubin less than or equal to 1.5 times ULN; aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 2.5 times ULN. For subjects with documented liver metastases, the AST/ALT may be less than or equal to 5 times ULN.
* Recovery to Grade 1 or baseline of any toxicity due to prior anticancer therapies (excluding alopecia).
* Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days prior to screening complete blood count (CBC) or Cycle 1, Day 1 treatment.
* Women of child bearing potential must have a negative serum pregnancy test.
* The effects of CUDC-907 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 30 days following the last study treatment.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

-Able to provide written informed consent and to follow protocol requirements.

EXCLUSION CRITERIA:

* Systemic anticancer therapy within 4 weeks of study entry, except for subjects with anaplastic/undifferentiated thyroid cancer who may be enrolled immediately after discontinuation of previous therapy.
* Other investigational agents within 4 weeks prior to study treatment except for subjects with anaplastic/undifferentiated thyroid cancer who may be enrolled immediately of discontinuation of previous therapy.
* Pregnant women are excluded from this study because the potential risk of teratogenic or abortifacient effects of CUDC-907 is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CUDC-907, breastfeeding should be discontinued if the mother is treated with CUDC-907. These potential risks may also apply to other agents used in this study.
* Diabetes mellitus that is not controlled with medication.
* Serious infection requiring intravenous antibiotic therapy within 14 days prior to study treatment.
* Evidence of central nervous system metastasis.
* Uncontrolled or severe cardiovascular disease, including myocardial infarction, unstable angina, or atrial fibrillation (AFib) within 6 months prior to study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, cardiac amyloidosis, or corrected QT interval (QTc) with Fridericia's (QTcF) correction that is unmeasurable or greater than or equal to 480 msec on screening electrocardiogram (ECG). (Note: for QTcF greater than or equal to 480 sec on the screening ECG, the ECG may be repeated twice at least 24 hours apart; the mean QTcF from the three screening ECGs must be < 480 msec in order to meet eligibility for trial participation).
* Gastrointestinal disease or disorder that could interfere with the swallowing, oral absorption, or tolerance of CUDC-907. This includes uncontrolled diarrhea (> 1 watery stool/day), major abdominal surgery, significant bowel obstruction and/or gastrointestinal diseases that could alter the assessment of pharmacokinetics or safety, including but not limited to: irritable bowel syndrome, ulcerative colitis, Crohn's disease and hemorrhagic coloproctitis.
* Unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a subject and/or compliance with the protocol.
* Second primary malignancy within 2 years of study entry other than adequately treated non-melanoma skin or superficial bladder cancer, curatively treated carcinoma in situ of the cervix or other curatively treated solid tumor deemed by the investigator to be at low risk for recurrence.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon D, Koehrle J, Reiners C, Boerner AR, Schmutzler C, Mainz K, Goretzki PE, Roeher HD. Redifferentiation therapy with retinoids: therapeutic option for advanced follicular and papillary thyroid carcinoma. World J Surg. 1998 Jun;22(6):569-74. doi: 10.1007/s002689900436. PMID 9597930
- [Background] Nilubol N, Kebebew E. Should small papillary thyroid cancer be observed? A population-based study. Cancer. 2015 Apr 1;121(7):1017-24. doi: 10.1002/cncr.29123. Epub 2014 Nov 25. PMID 25425528
- [Background] Kebebew E, Greenspan FS, Clark OH, Woeber KA, McMillan A. Anaplastic thyroid carcinoma. Treatment outcome and prognostic factors. Cancer. 2005 Apr 1;103(7):1330-5. doi: 10.1002/cncr.20936. PMID 15739211
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0029.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Anaplastic Thyroid Cancer: CUDC-907 for anaplastic thyroid cancer
  CUDC-907: 60 mg (2 capsules of 30 mg capsules) will be given orally once a day, 5 days on and 2 days off.
- Poorly Differentiated/Variants of Thyroid Cancer: CUDC-907 for Poorly differentiated and aggressive variants of differentiated thyroid cancer.
  CUDC-907: 60 mg (2 capsules of 30 mg capsules) will be given orally once a day, 5 days on and 2 days off.
Period: Overall Study
Arm/Group | Anaplastic Thyroid Cancer | Poorly Differentiated/Variants of Thyroid Cancer
Started | 4 | 3
Completed | 2 | 2
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaplastic Thyroid Cancer | Poorly Differentiated/Variants of Thyroid Cancer | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (19.18) | 66.6 (1.39) | 62.5 (16.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mexican, Puerto Rican, Cuban, Central/So American | 0 | 2 | 2
  Not meeting definition for Hispanic or Latino | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Response (Complete Response (CR) + Partial Response (PR)) Assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Clinical response, defined as a complete response + partial response (CR+PR) to CUDC-907 treatment, was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: Approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anaplastic Thyroid Cancer | Poorly Differentiated/Variants of Thyroid Cancer
Number analyzed (Participants) | 4 | 3
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

2. Secondary Outcome: Median Amount of Time Subject Survives Without Disease Progression After Treatment
Description: Time in days from initiation of treatment until tumor grows more than 20%. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or the appearance of one or more new lesions.
Time Frame: Approximately 6 months
Population: One participant was non-evaluable (withdrew consent).
Measure: Median (Full Range); unit: Days
Arm/Group | Anaplastic Thyroid Cancer | Poorly Differentiated/Variants of Thyroid Cancer
Number analyzed (Participants) | 3 | 2
Days | 31.3 [21 to 45] | 147 [127 to 167]

3. Secondary Outcome: Median Amount of Time Subject Survives After Therapy
Description: Time in days from the initiation of treatment until death estimated by the Kaplan-Meier method.
Time Frame: Approximately 12 months
Population: Participants are grouped together because of a small sample size and not enough power to compare the difference between two groups. No statistical analysis to be done.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- All Participants: CUDC-907 for anaplastic thyroid cancer CUDC-907: 60 mg (2 capsules of 30 mg capsules) will be given orally once a day, 5 days on and 2 days off.
  CUDC-907 for Poorly differentiated and aggressive variants of differentiated thyroid cancer.
  CUDC-907: 60 mg (2 capsules of 30 mg capsules) will be given orally once a day, 5 days on and 2 days off.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Days | 127 [66.5 to 187.5]

4. Secondary Outcome: Correlation Between Mutation Status of Tumor and Median Amount of Time Subject Survives Without Disease Progression After Treatment
Description: The amount of time subject survives without disease progression is compared by patient tumor mutation status.
Time Frame: At disease progression
Population: This outcome measure was not done. Data was collected but the correlation between mutation status of tumor and progression-free survival was not performed because of only BRAF V600E and the loss of tumor protein 53 (TP53) heterozygosity were found on a single patient each. Since only 1 mutant was found for each, no analysis was done.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation Between Activation of the Phosphoinositide 3-kinase (PI3K)/Protein Kinase B (AKT) and EGFR/RAS/RAF/MEK/ERK Pathways in Tumor Tissue and Median Amount of Time Subject Survives Without Disease Progression After Treatment
Description: The amount of time subject survives without disease progression is compared by the protein levels of PI3K/AKT and epidermal growth factor receptor (EGFR)/rat sarcoma (RAS)/rapidly accelerated fibrosarcoma (RAF)/methyl ethyl ketone (MEK)/extracellular-signal regulated kinase (ERK) in tumor tissue.
Time Frame: At disease progression
Population: This outcome measure was not done. Data was collected but no samples were analyzed because the experiment was not technically successful due to inconclusive results from immunohistochemistry (study of protein levels in tumor tissue) analysis of P13K/AKT and EGFR/RAS/RAF/MEK/ERK proteins.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation Between Histone Deacetylase 2 (HDAC2) and Survivin Protein Levels in Tumor Tissue With Median Amount of Time Subject Survives Without Disease Progression After Treatment
Description: The amount of time subject survives without disease progression is compared by the protein levels of HDAC2 and surviving in tumor tissue. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or the appearance of one or more new lesions.
Time Frame: At disease progression
Population: This outcome measure was not done. Data was collected but not analyzed because the assessment of HDAC2 and survivin proteins cannot be reliably performed with consistent results.
Groups:
- Anaplastic Cancer: CUDC-907 for anaplastic thyroid cancer CUDC-907: 60 mg (2 capsules of 30 mg capsules) will be given orally once a day, 5 days on and 2 days off.
Arm/Group | Anaplastic Cancer
Number analyzed (Participants) | 0

7. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 12 months and 13 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anaplastic Thyroid Cancer | Poorly Differentiated/Variants of Thyroid Cancer
Number analyzed (Participants) | 4 | 3
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 12 months and 13 days.
Arm/Group | Anaplastic Thyroid Cancer | Poorly Differentiated/Variants of Thyroid Cancer
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaplastic Thyroid Cancer (N=4) | Poorly Differentiated/Variants of Thyroid Cancer (N=3)
Death (General disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaplastic Thyroid Cancer (N=4) | Poorly Differentiated/Variants of Thyroid Cancer (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 4 (5) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03002623/Prot_SAP_ICF_000.pdf